CLINICAL TRIAL: NCT05483413
Title: Kütahya Health Science University
Brief Title: The Effect of Progressive Relaxation Exercises on Sleep Quality and Fatigue in Postmenopausal Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-41997688-050.99-34916
Record Dates: First submitted 2022-07-19; First posted 2022-08-02 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-06

CONDITIONS: Postmenopausal Period; Fatigue; Sleep Quality
Keywords: postmenopausal period; fatigue; sleep quality; progressive relaxation exercise
MeSH Terms: conditions — Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Relaxation Exercises (Experimental): Progressive relaxation exercises will be applied to this group for 8 weeks.
  Interventions: Behavioral: progressive relaxation exercises
- Standard of Care (No Intervention): This group will continue their routine coping habits against sleep and fatigue problems in the postmenopausal period for 8 weeks.

INTERVENTIONS:
Behavioral: progressive relaxation exercises — Progressive relaxation exercises are a cognitive behavioral technique that provides relaxation in the muscles that individuals can do alone.
  Arms: Progressive Relaxation Exercises

SUMMARY:
The population of the study will be postmenopausal women who applied to the KETEM unit of a hospital in western Turkey for examination. This study is a two-group randomized controlled study.

DETAILED DESCRIPTION:
The population of the study will be postmenopausal women who applied to the KETEM Unit of a hospital in western Turkey for examination. This study is a two-group randomized controlled study. These groups will be the experimental group to which Progressive Relaxation Exercises (PGE) will be applied and the control group who will continue their routine habits regarding sleep and fatigue problems in the postmenopausal period. Minimum number of women to be assigned to groups in the study; determined by power analysis.

To our knowledge, a sample size of 90 participants was selected and alpha=0.05 was selected to achieve 80% power to detect the traditionally moderate W=0.30 (moderate effect) differences between study groups, as we know of, according to the literature review. 1988; Foul et al, 2007). As a result, it was found that 60 women in total, 30 women in the experimental group and 30 women in the control group, should be included in the study. However, considering the risks such as women leaving the job over time and not being able to reach women, 3 women for each group (10% of the sample) will be included in the study as substitutes and it is anticipated that the research will be completed with a total of 66 women.

In order to provide an equal number of samples in the experimental and control groups and to ensure that both groups are similar in terms of all factors, except for the PGE application whose effectiveness will be examined, those who experience high levels of fatigue (high scores on the Piper Fatigue Scale) and low sleep quality (Pittsburg Sleep Quality Index) Randomization will be made between those who score 5 or more on the scales) and those who are similar in terms of independent variables. Randomizer.org program will be used to determine the women in the experimental and control groups, by choosing the "random randomization method" in order to provide an equal number of samples in both groups.

At the end of the randomization, difference analyzes will be made between the women who will be assigned to the experimental and control groups in terms of sociodemographic, menopausal and PGE-related characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Being in the postmenopausal period,
* Agreeing to participate in the research,
* Being able to read and write,
* Those experiencing high levels of fatigue
* Women with poor sleep quality

Exclusion Criteria:

* Experiencing menopause due to surgery, pharmacological reasons,
* Not being willing to participate in the study,
* Presence of any communication problems,
* Being in premenopause and perimenopause period.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Change in fatugue | 8-week process.
  At the end of 8 weeks of progressive relaxation exercises, change in fatigue
Change in sleep quality | 8-week process.
  At the end of 8 weeks of progressive relaxation exercises, change in sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Elif Tuğçe ÇİTİL, PhD, Study Director — Kütahya Health Science University
Locations (1):
- Kütahya Health Science University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided